CLINICAL TRIAL: NCT07234812
Title: The Effects of Tailored Resistance Exercise on Sleep Quality in Relation to Chronotype
Brief Title: Resistance Exercise and Sleep Quality by Chronotype
Acronym: TRE-SLEEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Aliaa Salem Mohamed Mohamed Menshawi, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: E-10840098-202.3.02-1592
Record Dates: First submitted 2025-09-23; First posted 2025-11-18 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Physical Therapy; Resistance Exercise; Sleep Disturbances; Sleep Quality; Chronotype; Circadian Rhythm; Health Behavior / Well-Being
Keywords: sleep disturbance; Sleep quality; Chronotype; Morningness-eveningness; Circadian rhythm; Resistance exercise; Home-based exercise; Sleep and exercise; Physical activity and sleep; Physical Therapy; Exercise; Telerehabilitation; Munich Chronotype Questionnaire (MCTQ); Pittsburgh Sleep Quality Index (PSQI); Mood (BRUMS, DASS-21); Randomized controlled trial; Physical therapy and rehabilitation
MeSH Terms: conditions — Parasomnias; Sleep Initiation and Maintenance Disorders; Health Behavior; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two parallel groups based on chronotype classification (morning type or evening type). Both groups will complete the same 8-week, moderate-intensity resistance exercise program delivered via online sessions three times per week in the morning. Outcomes will be compared between the two chronotype groups to evaluate whether the effects of exercise on sleep quality and mood differ by chronotype.
Masking Description: Participants will not be masked due to the nature of the supervised exercise sessions and chronotype classification. Outcome measures rely on self-reported questionnaires and standardized assessments, making blinding of participants impractical.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning Chronotype - Moderate-Intensity Resistance Exercise (Experimental): Participants identified as morning chronotypes (Munich Chronotype Questionnaire) will complete an 8-week, moderate-intensity resistance exercise program delivered online. Sessions are held in the morning, three times per week, lasting ~45 minutes (5-min warm-up, 35-min resistance training, 5-min cool-down). Exercises include push-ups, wall sits, squats, resistance band presses and pulls, rows, superman holds, and planks. Intensity is guided by 1RM testing, perceived exertion scales, and 7 point Likert scale of muscle soreness.
  Interventions: Behavioral: Moderate-Intensity Resistance Exercise Program
- Evening Chronotype - Moderate-Intensity Resistance Exercise (Experimental): Participants identified as evening chronotypes (Munich Chronotype Questionnaire) will complete an 8-week, moderate-intensity resistance exercise program delivered online. Sessions are held in the morning, three times per week, lasting ~45 minutes (5-min warm-up, 35-min resistance training, 5-min cool-down). Exercises include push-ups, wall sits, squats, resistance band presses and pulls, rows, superman holds, and planks. Intensity is guided by 1RM testing, perceived exertion scales, and 7 point Likert scale of muscle soreness.
  Interventions: Behavioral: Moderate-Intensity Resistance Exercise Program

INTERVENTIONS:
Behavioral: Moderate-Intensity Resistance Exercise Program — An 8-week, moderate-intensity resistance exercise program performed in the morning, 3 sessions/week on nonconsecutive days. Each 45-min session includes: 5-min warm-up (jumping jacks, high knees, running in place, hip hinge with reach, standing twists); 35-min progressive resistance training (Chest Press (Modified Push-Ups), Leg Press (Wall Sits with Squats), Squats, Shoulder Press (Resistance Band Overhead Press), Lat Pulldown (Resistance Band Pull-Downs), Rowing (Resistance Band Rows), Lower Back (Superman Holds), and Abdominals (Plank with Crunches)); and 5-min cool-down (Chest and Shoulder Stretch, Kneeling Hip Flexor Stretch, Standing Hamstring Stretch, Child's Pose with Side Stretch, and Cat-Cow Stretch ). Muscle soreness tracked after each session using 7-point Likert scale. Standardized videos, adherence checklists, resistance bands provided. Both chronotype groups complete identical sessions, outcomes compared.
  Other Names: Telerehabilitation Exercise; Resistance Training; Exercise Intervention; Strength Training

SUMMARY:
This study examines whether doing moderate resistance exercises in the morning can improve sleep quality and well-being in young adults. Participants with different daily activity patterns (morning or evening types) will take part in an 8-week online exercise program. The study will compare how exercise affects sleep, mood, and daily rhythm across these groups.

DETAILED DESCRIPTION:
Disturbed sleep is a widespread issue that affects health, mood, and daily function. Chronotype-the natural tendency to be active earlier or later in the day-may influence how people respond to exercise as a tool for improving sleep.

This trial investigates the effects of an 8-week, moderate-intensity resistance exercise program performed in the morning, delivered through telerehabilitation.

Participants include healthy young adults with self-identified morning or evening chronotypes. The study will measure changes in sleep quality, psychological well-being, alignment of daily rhythms, and will explore whether men and women respond differently to the program..

By comparing outcomes between chronotypes, this research aims to clarify whether exercise benefits are shaped by biological preference for morning or evening activity, or whether improvements occur regardless of chronotype.

The central question is whether improvements occur equally across chronotypes, or if biological preference shapes the response to exercise.

Null Hypothesis (H0): Moderate-intensity morning resistance exercise will have no differential effect on sleep quality, mood, or circadian alignment between participants with morning and evening chronotypes.

Alternative Hypothesis (H1):Moderate-intensity morning resistance exercise will have a differential effect on sleep quality, mood, or circadian alignment between participants with morning and evening chronotypes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 35 years
* Generally healthy, with mild to moderate sleep disturbance as categorized by the Pittsburgh Sleep Quality Index (PSQI)
* Body Mass Index (BMI) < 35 kg/m²
* No physical or organic limitations or diseases that would prevent participation in physical activity
* Non-smoker and non-alcoholic
* Caffeine consumption ≤ 2 cups per day (including coffee and energy drinks)
* Have not participated in more than 60 minutes/week of usual moderate-to-vigorous physical activity in the past 6 months, categorized as "moderate" on the International Physical Activity Questionnaire-Short Form (IPAQ-SF)
* No clinically diagnosed sleep apnea or other medical/psychiatric disorders responsible for sleep complaints
* Regular sleep schedule (no night shifts or transmeridian travel) in the 30 days prior to study enrollment
* Able to speak and write English

Exclusion Criteria:

* Current use of medications or psychotherapeutic drugs for insomnia or other psychiatric disorders
* Use of melatonin or other sleep aids in the past month
* Currently performing any aerobic or mind-body exercise classes (e.g., yoga, Pilates)
* Habitual daytime napping
* History of epilepsy or other convulsive disorders
* Pregnant individuals
* Habitual or recent use (within the past 30 days) of illegal drugs, psychotropic drugs, hypnotics, stimulants, or analgesics

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Sleep Quality Assessed by Pittsburgh Sleep Quality Index (PSQI) | Baseline, Week 4, and Week 8; primary comparison is change from baseline to Week 8
  Sleep quality will be measured using the Pittsburgh Sleep Quality Index (PSQI), a validated 19-item self-report questionnaire that evaluates sleep patterns over the past month. The PSQI generates seven component scores (subjective sleep quality, latency, duration, efficiency, disturbances, use of medication, daytime dysfunction), which are summed into a global score ranging from 0 to 21, with higher scores indicating poorer sleep quality. Assessments will be conducted at baseline (week 0), midpoint (week 4), and end of study (week 8). The primary endpoint is the change in global PSQI score from baseline to week 8, comparing differences between morning and evening chronotype groups following the resistance exercise program.

SECONDARY OUTCOMES:
Change in Circadian Alignment Assessed by Munich Chronotype Questionnaire (MCTQ) | Baseline and Week 8
  Chronotype and social jetlag will be evaluated using the MCTQ. The endpoint is change in chronotype alignment from baseline to week 8 and its relationship to exercise outcomes.
Change in Mood Assessed by Brunel Mood Scale (BRUMS) | Baseline, Week 4, and Week 8
  The Brunel Mood Scale (BRUMS) measures six mood states: anger, confusion, depression, fatigue, tension, and vigor. Higher scores reflect greater mood disturbance. Outcomes will track changes in mood from baseline to follow-up. It is a five-point Likert scale ranging from 0 (not at all) to 4 (extremely) according to their current feelings. The mood score is computed as the sum of all 24 items, with higher scores reflecting a greater intensity of that particular mood
Perceived Effort Assessed by OMNI Perceived Exertion Scale for Resistance Exercise (OMNI-RES) | Throughout Weeks 1-8
  The OMNI-RES is a 0-10 rating scale used to assess perceived exertion during resistance training. Higher scores reflect greater perceived effort. Participants will rate their exertion after each exercise session.
Muscle Soreness Assessed by 7-Point Likert Scale | After each exercise session, Weeks 1-8
  Participants will rate post-exercise soreness from 0 (no soreness) to 6 (severe soreness limiting movement) after each session to monitor tolerance.
Change in Physical Activity Level Assessed by International Physical Activity Questionnaire-Short Form (IPAQ-SF) | Baseline and Week 8
  The IPAQ-SF will measure weekly physical activity (MET-min/week and sedentary time). Outcomes include classification into low, moderate, or high activity.
Change in Mood Assessed by Depression Anxiety Stress Scales-21 (DASS-21) | Baseline, Week 4, and Week 8
  The DASS-21 is a 21-item questionnaire that evaluates symptoms of depression, anxiety, and stress. Higher scores indicate more severe symptoms. Outcomes will capture changes in psychological well-being across the intervention period. it is using a 4-point (0-3) Likert-type scale (ranging from "did not apply to me at all" 0, to "applied to me very much or most of the time" 3). Higher scores indicate greater severity of depression, anxiety, and stress symptoms, with subscale scores ranging from 0 to 42 and total scores from 0 to 126.
Change in Muscle Strength Assessed by One-Repetition Maximum (1RM) | Baseline, Week 4, and Week 8
  Muscle strength will be measured using the one-repetition maximum (1RM) test for selected resistance exercises. The primary outcome is change in maximal strength over the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Ergezen Şahin, Dr. Assistant Professor, Study Director — Department of Physiotherapy and Rehabilitation/Istanbul Medipol University
Locations (1):
- Medipol University, Istanbul, Beykoz/İstanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheville AL, Kollasch J, Vandenberg J, Shen T, Grothey A, Gamble G, Basford JR. A home-based exercise program to improve function, fatigue, and sleep quality in patients with Stage IV lung and colorectal cancer: a randomized controlled trial. J Pain Symptom Manage. 2013 May;45(5):811-21. doi: 10.1016/j.jpainsymman.2012.05.006. Epub 2012 Sep 24. PMID 23017624
- [Background] Karandikar-Agashe G, Agrawal R. Comparative Study of the Effect of Resistance Exercises versus Aerobic Exercises in Postmenopausal Women Suffering from Insomnia. J Midlife Health. 2020 Jan-Mar;11(1):2-5. doi: 10.4103/jmh.JMH_35_19. Epub 2020 May 4. PMID 32684719
- [Background] Passos GS, Poyares D, Santana MG, Garbuio SA, Tufik S, Mello MT. Effect of acute physical exercise on patients with chronic primary insomnia. J Clin Sleep Med. 2010 Jun 15;6(3):270-5. PMID 20572421
- [Background] de Sa Souza H, de Melo CM, Piovezan RD, Miranda REEPC, Carneiro-Junior MA, Silva BM, Thomatieli-Santos RV, Tufik S, Poyares D, D'Almeida V. Resistance Training Improves Sleep and Anti-Inflammatory Parameters in Sarcopenic Older Adults: A Randomized Controlled Trial. Int J Environ Res Public Health. 2022 Dec 6;19(23):16322. doi: 10.3390/ijerph192316322. PMID 36498393
- [Background] Maric D, Ficarra S, Di Bartolo L, Rossi C, Asimakopoulou Z, Vantarakis A, Carbonell-Baeza A, Jimenez-Pavon D, Gomes B, Tavares P, Baxter R, Pusa S, Thaller P, Papakonstantinou S, Kirkar M, Glorioso F, Galioto M, Gentile A, Thomas E, Bianco A. Effects of resistance training on sleep quality and disorders among individuals diagnosed with cancer: A systematic review and meta-analysis of randomized controlled trials. Cancer Med. 2024 Apr;13(8):e7179. doi: 10.1002/cam4.7179. PMID 38650577
- [Background] Vickers AJ. Time course of muscle soreness following different types of exercise. BMC Musculoskelet Disord. 2001;2:5. doi: 10.1186/1471-2474-2-5. Epub 2001 Oct 23. PMID 11701094
- [Background] Morishita S, Tsubaki A, Takabayashi T, Fu JB. Relationship between the rating of perceived exertion scale and the load intensity of resistance training. Strength Cond J. 2018 Apr;40(2):94-109. doi: 10.1519/SSC.0000000000000373. PMID 29674945
- [Background] Robertson RJ, Goss FL, Rutkowski J, Lenz B, Dixon C, Timmer J, Frazee K, Dube J, Andreacci J. Concurrent validation of the OMNI perceived exertion scale for resistance exercise. Med Sci Sports Exerc. 2003 Feb;35(2):333-41. doi: 10.1249/01.MSS.0000048831.15016.2A. PMID 12569225
- [Background] Terry PC, Lane AM, Lane HJ, Keohane L. Development and validation of a mood measure for adolescents. J Sports Sci. 1999 Nov;17(11):861-72. doi: 10.1080/026404199365425. PMID 10585166
- [Background] Carney CE, Buysse DJ, Ancoli-Israel S, Edinger JD, Krystal AD, Lichstein KL, Morin CM. The consensus sleep diary: standardizing prospective sleep self-monitoring. Sleep. 2012 Feb 1;35(2):287-302. doi: 10.5665/sleep.1642. PMID 22294820
- [Background] Seo DI, Kim E, Fahs CA, Rossow L, Young K, Ferguson SL, Thiebaud R, Sherk VD, Loenneke JP, Kim D, Lee MK, Choi KH, Bemben DA, Bemben MG, So WY. Reliability of the one-repetition maximum test based on muscle group and gender. J Sports Sci Med. 2012 Jun 1;11(2):221-5. eCollection 2012. PMID 24149193
- [Background] Sjostrom, M., Ainsworth, B.E., Bauman, A., Bull, F.C., Hamilton-Craig, C.R., & Sallis, J.F. (2005). Guidelines for data processing analysis of the International Physical Activity Questionnaire (IPAQ) - Short and long forms.
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Zavada A, Gordijn MC, Beersma DG, Daan S, Roenneberg T. Comparison of the Munich Chronotype Questionnaire with the Horne-Ostberg's Morningness-Eveningness Score. Chronobiol Int. 2005;22(2):267-78. doi: 10.1081/cbi-200053536. PMID 16021843
- [Background] Kantermann T, Sung H, Burgess HJ. Comparing the Morningness-Eveningness Questionnaire and Munich ChronoType Questionnaire to the Dim Light Melatonin Onset. J Biol Rhythms. 2015 Oct;30(5):449-53. doi: 10.1177/0748730415597520. Epub 2015 Aug 4. PMID 26243627
- [Background] Kim N, Ka S, Park J. Effects of exercise timing and intensity on physiological circadian rhythm and sleep quality: a systematic review. Phys Act Nutr. 2023 Sep;27(3):52-63. doi: 10.20463/pan.2023.0029. Epub 2023 Sep 30. PMID 37946447
- [Background] Ferris LT, Williams JS, Shen CL, O'Keefe KA, Hale KB. Resistance training improves sleep quality in older adults a pilot study. J Sports Sci Med. 2005 Sep 1;4(3):354-60. eCollection 2005 Sep 1. PMID 24453540
- [Background] Flausino NH, Da Silva Prado JM, de Queiroz SS, Tufik S, de Mello MT. Physical exercise performed before bedtime improves the sleep pattern of healthy young good sleepers. Psychophysiology. 2012 Feb;49(2):186-92. doi: 10.1111/j.1469-8986.2011.01300.x. Epub 2011 Oct 6. PMID 22092095
- [Background] Kredlow MA, Capozzoli MC, Hearon BA, Calkins AW, Otto MW. The effects of physical activity on sleep: a meta-analytic review. J Behav Med. 2015 Jun;38(3):427-49. doi: 10.1007/s10865-015-9617-6. Epub 2015 Jan 18. PMID 25596964
- [Background] Institute of Medicine (US) Committee on Sleep Medicine and Research; Colten HR, Altevogt BM, editors. Sleep Disorders and Sleep Deprivation: An Unmet Public Health Problem. Washington (DC): National Academies Press (US); 2006. Available from http://www.ncbi.nlm.nih.gov/books/NBK19960/ PMID 20669438
- See also: National Sleep Foundation's sleep time duration recommendations: methodology and results summary — https://doi.org/10.1016/j.sleh.2014.12.010
- See also: Effects of resistance exercise training and stretching on chronic insomnia — https://doi.org/10.1590/1516-4446-2018-0030
- See also: Resistance training improves sleep quality, redox balance and inflammatory profile in maintenance hemodialysis patients: a randomized controlled trial. — https://doi.org/10.1038/s41598-020-68602-1